CLINICAL TRIAL: NCT06000176
Title: Comparison of Optical Coherence Tomography Angiography Microvascular Changes in Primary Open Angle and Primary Angle Closure Glaucoma
Status: Completed | Type: Observational
Sponsor: Omar Said (Other)
Responsible Party: Sponsor-Investigator, Omar Said, Assistant Professor Of Ophthalmology, Fayoum University
Organization: Fayoum University (Other)
Other Study IDs: M557
Record Dates: First submitted 2023-08-12; First posted 2023-08-21 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Glaucoma,Primary Open-Angle ,Primary Angle Closure
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- interventional details : diagnostic test OCTA macula and ONH: interventional details : diagnostic test OCTA macula and ONH in the 3 groups
  Interventions: Device: Optical coherence tomography angiography

INTERVENTIONS:
Device: Optical coherence tomography angiography — diagnostic test OCTA macula and ONH

SUMMARY:
This work aims to study the peripapillary and macular microvascular changes in primary open angle and primary angle closure glaucoma using Optical Coherence Tomography Angiography (OCTA).

DETAILED DESCRIPTION:
After approval of the local institutional ethics committee and local institutional review board, all patients presenting to the outpatient clinic of the department of Ophthalmology in the universities has been subjected to routine ophthalmological examination including: best corrected visual acuity (BCVA), Slit-lamp evaluation of anterior segment, IOP by Goldmann applanation tonometer, Gonioscopy using gonio contact lens, Fundus examination by indirect opthalmoscope with history taking focusing on positive family history of glaucoma after a detailed informed consent was signed by eligible patients and investigated by OCTA of the Peripapillary and Macular vascular density on presentation using AngiVue (Optovue, Inc., Fremont, CA, USA).

Data analysis performed using the Statistical Package of Social Science (SPSS) software version 22 in windows 7 (SPSS Inc., Chicago, IL, USA) Simple descriptive statistical analysis in the form of numbers and percentages of qualitative data, and arithmetic means as central tendency measurement, standard deviations as a measure of dispersion of quantitative parametric data.

For quantitative parametric data: Independent samples test was used to compare quantitative measures between two independent groups, One-way analysis of variance ANOVA test used to compare quantitative measures between more than two independent groups of quantitative data with the benferroni Post-HOC to test the significance between each two groups, Paired t-test used to compare two dependent quantitative data.

For qualitative data Chi square test used to compare between two or more than two qualitative groups.

Bivariate Pearson correlation test to test the association between variables The probability value (P-value) < 0.05 was considered as statistical significant

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old.
* Fulfilling Diagnostic criteria of PACG patients :occluded angle by gonioscopy in which > 180˚ of trabecular meshwork cannot be seen , IOP>21, Optic disc and RNFL damage due to glaucoma
* Diagnosed POAG patient: open anterior chamber angle ,IOP>21 ,Optic disc and RNFL damage due to glaucoma
* Healthy patient: normal anterior chamber, open angle and normal fundus.

Exclusion Criteria:

* History of other causes of optic neuropathy.
* History of systemic diseases. (HTN, DM, Cardiac).
* Previous ocular surgeries or Laser iridotomy.
* Poor quality of OCTA image less than 4/10.
* Refractive errors > 6 diopters sphere, >3 diopter cylinder
* Poor cooperation or fixation with the OCTA examination.
* Secondary causes of glaucoma
* Media opacity that interfere with quality of image (dense cataract,corneal opacity,…)
* Previous acute attack of ACG

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with primary open angle ,primary angle closure glaucoma and control patients
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2022-04-05 (Actual); Primary Completion 2023-07-20 (Actual); Study Completion 2023-07-20 (Actual)

PRIMARY OUTCOMES:
OCTA macula and ONH | We will recruit patient that include the inclusion criteria from april2022 to july 2023
  macular 6*6,3*3 and peripapillary vessel density

CONTACTS AND LOCATIONS:
Locations (1):
- Athar Mohamed Mohamed Makhlouf, Al Fayyum, Egypt

IPD SHARING:
Plan to Share IPD: Undecided